CLINICAL TRIAL: NCT01878799
Title: An Open Label Trial to Assess Safety, Tolerability, and Efficacy of the Fixed Dose Combination of GS-7977 and GS-5885 in HCV Genotype 1 Subjects Coinfected With HIV
Brief Title: Study of A Combination Pill With GS-7977 and GS-5885 for Hepatitis C in People With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130159; 13-I-0159
Record Dates: First submitted 2013-06-14; First posted 2013-06-17 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C; HIV
Keywords: Direct Acting Antiviral; Treatment Naive; Interferon Sparing; Ribavirin Sparing
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV (Experimental): Subjects with HIV and HCV
  Interventions: Drug: GS-7977/GS- 5885 FDC

INTERVENTIONS:
Drug: GS-7977/GS- 5885 FDC — The GS-7977/GS-5885 FDC product combines a potent HCV nucleotide inhibitor and a potent HCV NS5A inhibitor and will be given for 12 weeks.

SUMMARY:
Background:

- Present treatment for hepatitis C includes the use of a weekly injection and two different pills. This treatment is associated with serious side effects. Drugs that can be taken by mouth and cure HCV infection without serious side effects would be a great help to the large number of people infected with HCV. GS-7977 and GS-5885 are new medications being developed to treat the hepatitis C virus (HCV) infection. They are still being researched and are not approved by the Food and Drug Administration. They are being developed as treatment for hepatitis C as a single pill taken once a day.

Objectives:

- To determine whether a combination of the two study drugs can safely and effectively treat HCV infection in people with HIV infection and who do not have cirrhosis of the liver.

Eligibility:

- Individuals who have HIV infection and have liver disease caused by infection with HCV.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Urine samples will be collected from participants who might become pregnant. If a participant has not had a liver biopsy in the past 3 years, one will be required.
* Participants will take one pill daily for 12 weeks. This pill will be a combination of the two study drugs.
* Treatment will be monitored with frequent clinic visits and blood tests over a total of 60 weeks.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the US an estimated 4.1 million people are infected with HCV which is the principal cause of death from liver disease and leading indication for liver transplantation. Significant advances have been made with the approval of directly acting antivirals (DAA) namely the protease inhibitors, telaprevir (TVR) and boceprevir (BOC) which have been shown to significantly improve rates of sustained virologic response (SVR). Response rates to these new combinations in HIV/HCV are also very promising, however treatment has been characterized with high rates of toxicities.

Recently several trials have confirmed the efficacy of potent DAA therapy without concomitant IFN in the treatment of HCV monoinfected individuals. Given the improved response rates achieved with a combination of DAAs with fast HCV suppression and improved side-effect profiles; and the need for better therapy for HIV/HCV co-infected subjects, we propose a study to determine the safety, tolerability and efficacy of 12 weeks of treatment with a fixed dose combination of GS-7977 and GS-5885 in HIV/HCV Genotype 1 (GT-1) subjects. We hypothesize that anti-HCV therapy that does not rely on the host immune system will provide an enhanced rate of SVR among HIV/HCV GT-1 coinfected subjects. The findings from this study will aid in our understanding of determinants of response to an IFN-free regimen in HIV/HCV coinfected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Eighteen years of age or older at screening.
  2. HCV treatment-naive, as defined as no prior exposure to any IFN, RBV, or other approved or experimental HCV-specific direct-acting antiviral agent.
  3. Participants must be willing to practice either:

     1. Abstinence from sexual intercourse or
     2. At least 2 forms of contraception including one barrier method from 2 weeks prior to Day 0 through 30 days after the last dose is received.

     i. Female partners of male study subjects may rely upon hormonal contraception as one of the 2 methods; however female study subjects may not.
  4. Chronic hepatitis C infection defined as one of the following:

     1. Positive for anti-HCV antibody, HCV RNA, or an HCV genotype at least 6 months before screening, and positive for HCV RNA and anti-HCV antibody at the time of screening or
     2. Positive for anti-HCV antibody and HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of chronic hepatitis C disease, such as the presence of fibrosis).
  5. HIV treatment status:

     1. Documented HIV infection, ARV untreated for > 8 weeks preceding dosing and having either:

        1. a CD4 T-cell count greater than or equal to 500 cells/mm3 within 8 weeks of Day 0 or
        2. an HIV viral load less than 500 copies/mL with a stable CD4 count for at least 3 months.
     2. Documented HIV infection on a stable, protocol-approved, ARV regimen for greater than or equal to 8 weeks prior to dosing and is expected to continue the current ARV regimen through the end of study with all of the following:

        1. a CD4 T-cell count > 100 cells/mm3
        2. a documented plasma HIV-1 RNA level less than the level of detection for at least 8 weeks preceding dosing.

           If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL (e.g.,< 20 copies/mL), the Screening plasma HIV-1 RNA level cannot exceed 50 copies/mL.
        3. HIV ARV agents including only combination regimens consisting of medications from the following list: tenofovir (TDF), emtricitabine (FTC), efavirenz, raltegravir, and rilpivirine administered according to their manufacturer s prescribing information. (reference Section 10.3 for additional information)
  6. Documentation of hepatitis C genotype 1a, 1b or mixed 1a/1b
  7. Absence of cirrhosis, defined as one of the following:

     1. A liver biopsy performed within 36 calendar months of screening showing absence of cirrhosis.
     2. FibroTest score of < 0.48 AND APRI of < 1 performed during the 8 weeks preceding dosing (In the absence of a definitive diagnosis of presence or absence of cirrhosis by the above criteria, a liver biopsy is required).
  8. Able to effectively communicate with the Investigator and other center personnel.
  9. Willing to give written informed consent and comply with the study restrictions and requirements.
  10. If opioid-dependent, subjects must be participating in a supervised treatment.
  11. Participants must have a primary medical provider outside of OP8 and the NIH for medical management.

EXCLUSION CRITERIA:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Current or prior history of any of the following:

   1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
   2. Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
   3. Poor venous access interfering with required study blood collection.
   4. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
   5. Solid organ transplantation.
   6. Significant pulmonary disease, significant cardiac disease or porphyria.
   7. Unstable psychiatric disease (Subjects with psychiatric illness that is well-controlled on a stable treatment regimen or currently not requiring medication may be included).
   8. Any malignancy or its treatment that in the opinion of the PI may cause ongoing interference with host immunity; subjects under evaluation for malignancy are not eligible.
   9. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
   10. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson s disease, alfa-1 antitrypsin deficiency, cholangitis).
   11. Patients with renal impairment or uncontrolled medical problems that could place them at high risk for developing renal impairment.
2. Positive test at screening for either HBsAg or quantifiable HBV DNA (completed only if necessary to rule out chronic HBV)
3. Current use of non-protocol approved ARVs.
4. A new AIDS-defining condition diagnosed within 30 days prior to screening or active, serious infection (other than HIV or HCV) requiring parenteral antibiotics, antivirals or antifungals within 30 days prior to Day 0.
5. Cirrhosis of the liver
6. Screening or baseline ECG with clinically significant ECG findings.
7. Abnormal hematological and biochemical parameters, including:

   1. Neutrophil count < 750 cells/mm(3)
   2. Hemoglobin < 9 g/dL. If Hgb is < 11g/dL in women or < 12 g/dL in men. Other causes of anemia should be excluded as medically indicated.
   3. Platelet count less than or equal to 50,000 cells/mm(3)
   4. Estimated GFR (calculated by the CKD-EP(I) equation) < 50 mL/min/per 1.73 m(2) if not on ARV or < 60 mL/min if on ARVs
   5. ALT or AST greater than or equal to 10 times ULN
   6. Serum lipase greater than or equal to 1.5 times ULN (at screening or during the screening period)
   7. Direct bilirubin greater than or equal to 1.50 times ULN
   8. Albumin less than or equal to 3.0 g/dL
   9. INR greater than or equal to 1.5 times ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
8. Donation or loss of more than 400 mL blood within 8 weeks prior to first dose administration.
9. Poorly controlled diabetes mellitus indicated by hemoglobin A1C > 10% at screening for known diabetics.
10. Known hypersensitivity to, GS-5885, GS-7977, or formulation excipients.
11. Pregnant/Breastfeeding women.
12. Co-enrollment in other clinical trials is restricted, and requires approval of the Investigator.

    Study staff should be notified of co-enrollment status.
13. Need for use of the following medications from 21 days prior to the start of study drugs through the end of treatment:

    1. Hematologic stimulating agents (e.g. erythropoiesis-stimulating agents (ESAs); granulocyte colony stimulating factor (GCSF); thrombopoietin (TPO) mimetics)
    2. Chronic systemic immunosuppressants including, but not limited to, corticosteroids (prednisone equivalent of > 10 mg/day for > 2 weeks), azathioprine, or monoclonal antibodies (e.g., infliximab)
    3. Investigational agents or devices for any indication
    4. Medications for disease conditions excluded from the protocol (e.g., active cancer, transplantation) are not listed under this Concomitant Medication section and are disallowed in the study.
    5. Concomitant use of certain medications or herbal/natural supplements per PI discretion expected to result in pharmacokinetic interactions resulting in increases or decreases in exposure of study drug(s) as listed in Table of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kottilil, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Kim WR. The burden of hepatitis C in the United States. Hepatology. 2002 Nov;36(5 Suppl 1):S30-4. doi: 10.1053/jhep.2002.36791. PMID 12407574
- [Derived] Townsend K, Petersen T, Gordon LA, Kohli A, Nelson A, Seamon C, Gross C, Tang L, Osinusi A, Polis MA, Masur H, Kottilil S. Effect of HIV co-infection on adherence to a 12-week regimen of hepatitis C virus therapy with ledipasvir and sofosbuvir. AIDS. 2016 Jan;30(2):261-6. doi: 10.1097/QAD.0000000000000903. PMID 26691547
- [Derived] Osinusi A, Townsend K, Kohli A, Nelson A, Seamon C, Meissner EG, Bon D, Silk R, Gross C, Price A, Sajadi M, Sidharthan S, Sims Z, Herrmann E, Hogan J, Teferi G, Talwani R, Proschan M, Jenkins V, Kleiner DE, Wood BJ, Subramanian GM, Pang PS, McHutchison JG, Polis MA, Fauci AS, Masur H, Kottilil S. Virologic response following combined ledipasvir and sofosbuvir administration in patients with HCV genotype 1 and HIV co-infection. JAMA. 2015 Mar 24-31;313(12):1232-9. doi: 10.1001/jama.2015.1373. PMID 25706232

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With HIV and HCV on Antiretroviral Agents: Subjects with HIV and HCV on antiretroviral agents given 'Drug: GS-7977 (sofosbuvir 400mg)/GS-5885 (ledipasvir 90mg) FDC' once daily by mouth for 12 weeks. The GS-7977/GS-5885 product combines a potent HCV nucleotide inhibitor and a potent HCV NS5A inhibitor.
- Subjects With HIV and HCV Who Are Not on Antiretroviral Agents: Subjects with HIV and HCV not on antiretroviral agents given 'Drug: GS-7977 (sofosbuvir 400mg)/GS-5885 (ledipasvir 90mg) FDC' once daily by mouth for 12 weeks. The GS-7977/GS-5885 product combines a potent HCV nucleotide inhibitor and a potent HCV NS5A inhibitor.
Period: Overall Study
Arm/Group | Subjects With HIV and HCV on Antiretroviral Agents | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents
Started | 37 | 13
Completed | 36 | 13
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With HIV and HCV Who Are Not on Antiretroviral Agents: Subjects with HIV and HCV who are not on antiretroviral agents given 'Drug: GS-7977 (sofosbuvir 400mg)/GS-5885 (ledipasvir 90mg) FDC' once daily by mouth for 12 weeks. The GS-7977/GS-5885 product combines a potent HCV nucleotide inhibitor and a potent HCV NS5A inhibitor.
- Total: Total of all reporting groups
Arm/Group | Subjects With HIV and HCV on Antiretroviral Agents | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents | Total
Number analyzed (Participants) | 37 | 13 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 13 | 45
  >=65 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 30 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 13 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 10 | 41
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Achieved SVR12 (HCV RNA <LLOQ 12 Weeks After Completion of Treatment)
Description: The primary end point was sustained virologic response [plasma HCV RNA level <12 IU/mL by real-time HCV assay (Abbott)] at 12 weeks after treatment completion (SVR12) among all patients enrolled in the study.
Time Frame: 12 weeks after completion of treatment
Population: The analysis included all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subjects With HIV and HCV on Antiretroviral Agents | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents
Number analyzed (Participants) | 37 | 13
percentage of participants | 97 [89 to 100] | 100 [75 to 100]

ADVERSE EVENTS:
Time Frame: On or after the first dose of the study drug up to date of last dose of study drug (12 weeks) plus 30 days
Arm/Group | Subjects With HIV and HCV on Antiretroviral Agents | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/13
Other Adverse Events (participants affected / at risk) | 36/37 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With HIV and HCV on Antiretroviral Agents (N=37) | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents (N=13)
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With HIV and HCV on Antiretroviral Agents (N=37) | Subjects With HIV and HCV Who Are Not on Antiretroviral Agents (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
Pain (General disorders) | 2 | 3
Seasonal allergy (Immune system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 2
Amylase increased (Investigations) | 13 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 0
Blood bicarbonate abnormal (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood cholesterol increased (Investigations) | 16 | 5
Blood creatinine increased (Investigations) | 6 | 0
Hemoglobin decreased (Investigations) | 4 | 0
Lipase increased (Investigations) | 5 | 0
Low density lipoprotein increased (Investigations) | 9 | 3
Neutrophil count decreased (Investigations) | 8 | 5
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 9
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Hypoesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Bereavement (Social circumstances) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes